CLINICAL TRIAL: NCT05715723
Title: Non-interventional, Prospective Study of Safety and Efficiency of the Drug Reamberin® in the Intensive Care of Patients With Acute Ethanol Intoxication: Hospital Practice
Brief Title: Study of Safety and Efficiency of the Drug Reamberin® in the Intensive Care of Patients With Acute Ethanol Intoxication
Status: Completed | Type: Observational
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Other Study IDs: Reamberin\2022\01
Record Dates: First submitted 2022-12-28; First posted 2023-02-08 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2024-11

CONDITIONS: Ethanol Intoxication
Keywords: reamberin; intensive care; acute ethanol intoxication; Ethanol Intoxication
MeSH Terms: interventions — Reamberin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The control group: Standard therapy
- The test group: Standard therapy + Reamberin
  Interventions: Drug: Reamberin

INTERVENTIONS:
Drug: Reamberin — Reamberin® in the average daily dose of 10 ml/kg daily
  Groups: The test group

SUMMARY:
Acute ethanol intoxication is the most frequent pathologic condition developing in subjects using alcohol. The severity of disorders in acute alcohol intoxication is determined, first of all, by the quantity of consumed alcohol and the duration of the toxic effect. When toxic doses of alcohol are taken per os, a life-threatening condition develops, which is manifested by consciousness depression and severe metabolism disorders. Reamberin (1.5 % meglumine sodium succinate solution) is an infusion solution with a balanced electrolyte composition and succinic acid, which is recommended for rehydration and detoxication in patients with intoxications of different genesis. The metabolic effect of Reamberin helps restore homeostasis and improve the natural organism detoxication. The investigators suppose that administration of Reamberin to patients with acute ethanol intoxication will make it possible to improve the treatment quality as compared to the standard therapy.

DETAILED DESCRIPTION:
All drugs will be administered according to the instruction for medical use and conventional clinical practice.

The decision on the selection of therapy shall be made by a medical investigator irrespective of the protocol before the inclusion of a patient in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged from 22 to 65 years.
2. It is planned to administer one of the following treatment types to the patient, as part of the routine clinical practice:

   * Standard fluid administration + Reamberin®. It is planned to administer the drug Reamberin® in the average daily dose of 10 ml/kg daily for the whole period of treatment at ICU.
   * Standard fluid administration (without the use of the drug Reamberin®).
3. Primary diagnosis:

   * toxic effect of ethanol (T51.0 according to ICD-10);
   * acute intoxication caused by the simultaneous use of several narcotic drugs and the use of other psychoactive substances2 (F19.0 according to ICD-10);
   * mental and behavioral disorders caused by alcohol use. Acute intoxication (F10.0 according to ICD-10).
4. Blood ethanol concentration: 1.5 ‰ (per mille) and more.
5. Consciousness depression (Glasgow Coma Score = 6-12)
6. Laboratory signs of a shift in the acid-base balance towards metabolic acidosis: base deficit (BE) of venous blood less than -2.2 mmol/l).
7. Availability of the written consent of the patient or his (her) legally authorized representative.

Exclusion Criteria:

1. Use of other drugs containing malate or succinate.
2. Consciousness depression with Glasgow Coma Score of lower than 6.
3. Intoxication with addictive substances and psychotropic drugs.
4. Shock.
5. Body weight of less than 50 kg or more than 120 kg.
6. Data on the presence of malignant neoplasms.
7. Decompensation of chronic pulmonary diseases with the development of respiratory failure of degree II-III as at the time of inclusion in the study.
8. Pregnancy, breast feeding.
9. Craniocerebral injury or polytrauma.
10. Acute cerebrovascular accident.
11. Infection-inflammatory disease of CNS (meningitis, encephalitis etc.) and other variants of CNS function disorder not associated with ethanol intoxication.
12. Respiratory impairment requiring ALV.
13. Contraindications mentioned in the approved instructions for the use of the drugs used in the study.
14. A disease or the use of drugs, which, in the physician's opinion, can influence safety, tolerance and efficiency of the study drugs.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ethanol intoxication, hospitalized to an intensive care unit with signs of toxic encephalopathy (consciousness depression level: Glasgow Coma Score = 6-12) and metabolic acidosis
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Difference in the average stay duration at ICU between patient groups. | Up to 2 weeks
Difference in the average consciousness recovery duration between patient groups. | Up to 2 weeks

SECONDARY OUTCOMES:
Difference in average blood lactate levels between the groups, measured at the baseline and after 24 hours of the therapy | Baseline, 24 hours after the intervention
Difference in average serum bicarbonate levels between the groups, measured at the baseline and after 24 hours of the therapy | Baseline, 24 hours after the intervention
Percentage of patients, whose consciousness recovered to Glasgow Coma Score of up to 14 after 24 hours of the therapy, measured in both groups. | 24 hours after the intervention
  The Glasgow Coma Scale: 15 points - clear consciousness.
  14-13 points - moderate stunning.
  12-11 points - deep stunning.
  10-8 points - sopor.
  7-6 points - moderate coma.
  5-4 points - deep coma.
  3 points - terminal coma, brain death.
Dynamics of serum bicarbonate levels during the study (at the baseline, in 24 hours, by the end of the treatment in ICU), measured in both groups. | Baseline, 24 hours after the intervention, up to 2 weeks
Dynamics of organ failure score according to SOFA scale during the study, measured in both groups. | Baseline, 24 hours after the intervention, up to 2 weeks
  Sepsis-related Organ Failure scale: min 0 points, max 24 points. The higher the total score, the higher the degree of multiple organ failure
Dynamics of consciousness level score according to Glasgow Coma Scale during the study, measured in both groups. | Baseline, 24 hours after the intervention, up to 2 weeks
  The Glasgow Coma Scale: 15 points - clear consciousness.
  14-13 points - moderate stunning.
  12-11 points - deep stunning.
  10-8 points - sopor.
  7-6 points - moderate coma.
  5-4 points - deep coma.
  3 points - terminal coma, brain death.
Dynamics of the total score according to ICDSC scale (Intensive Care Delirium Screening Checklist) during the study, measured in both groups | Baseline, 24 hours after the intervention, up to 2 weeks
  Intensive Care Delirium Screening Checklist: ыcore ≥ 4 - delirium
Percentage of patients, who developed delirium, measured in both groups | Up to 2 weeks
Percentage of patients, who developed hospital-acquired pneumonia, measured in both groups | Up to 2 weeks
Percentage of patients, who developed extrapulmonary complications, measured in both groups. | Up to 2 weeks
Percentage of lethal outcomes for the whole study period, measured in both groups. | Up to 2 weeks
Percentage of patients, for whom it became necessary to administer ALV, over the whole study period, measured in both groups. | Up to 2 weeks

CONTACTS AND LOCATIONS:
Locations (18):
- Russia (18):
  - City Clinical Hospital of Emergency Medical Care, Kaliningrad
  - K.N. Shevchenko Kaluga Regional Clinical Hospital of Emergency Medical Care, Kaluga
  - M.A. Podgorbunsky Kuzbass Clinical Hospital of Emergency Medical Care, Kuzbass
  - Buyanov City Clinical Hospital, Moscow
  - KORSAKOV Medical Center, Moscow
  - N.V. Sklifosovsky Research Institute of Emergency Care of the Moscow City Health Department, Moscow
  - Negovsky Research Institute of General Intensive Care Medicine, Moscow
  - Zhukovskaya City Clinical Hospital, Moscow
  - City Clinical Hospital No. 2, Novosibirsk
  - City Clinical Hospital of Emergency Medicine No. 1, Omsk
  - Regional Clinical Hospital,, Ryazan
  - City Mariinskaya Hospital, Saint Petersburg
  - City Narcological Hospital, Saint Petersburg
  - Dzhanelidze St. Petersburg Research Institute of Emergency Medicine, Saint Petersburg
  - State Healthcare Institution Saratov Yu. Ya. Gordeev City Clinical Hospital No. 1, Saratov
  - V.N. Koshelev City Clinical Hospital No. 6, Saratov
  - Tyumen State Medical University, Tyumen
  - Yaroslavl Regional Clinical Narcological Hospital, Yaroslavl

IPD SHARING:
Plan to Share IPD: No